CLINICAL TRIAL: NCT06073873
Title: Post-Marketing Surveillance (PMS) Study on Zeposia® (Ozanimod) Use Among Moderate to Severe Active Ulcerative Colitis Patients in Korea
Brief Title: A Post-Marketing Surveillance Study to Assess Safety of Ozanimod in Patients With Moderate to Severe Active UC in Korea
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM047-024
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ozanimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with moderate to severe active ulcerative colitis treated with ozanimod
  Interventions: Drug: Ozanimod

INTERVENTIONS:
Drug: Ozanimod — According to local product label

SUMMARY:
The purpose of this observational study is to assess the real-world safety of ozanimod in Korean participants with moderate to severe active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants 19 years of age or older
* Participants who will receive ozanimod according to the approved label after enrollment
* Participants who sign the informed consent form voluntarily

Exclusion Criteria:

* Participants who are prescribed ozanimod for therapeutic indications not approved in Korea
* Participants for whom ozanimod is contraindicated as clarified in Korean prescribing information approved by Ministry of Food and Drug Safety

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of participants with moderately to severely active ulcerative colitis who will receive at least 1 dose of ozanimod according to local product label. Moderate to severe disease will be defined as a Mayo score of 6 to 12 and an endoscopic sub-score of 2 or higher. Participants will be eligible if they had an inadequate response, lost response, or were intolerant to conventional therapy (5-aminosalicylic acid, corticosteroids, immunosuppressants) or biologic agents.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Up to 52 weeks
  The type, frequency, seriousness and severity of adverse events (AEs), and relationship of AEs for ozanimod

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol-Myers Squibb YH, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts